CLINICAL TRIAL: NCT06256406
Title: Comparative Evaluation Between Preterms and Newborns Undergoing Surgery. Effectiveness of a Multimodal Sensory Intervention on Newborns and Parents' Stress
Brief Title: Effects of Confortable Environment, Kangaroo Care and Music Therapy in Newborns in Neonatal Intensive Care Unit
Acronym: PRE-CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Universitario, Catania (Other)
Responsible Party: Principal Investigator, Pasqua Betta, Principal investigator, Policlinico Universitario, Catania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 122/2022/PO
Record Dates: First submitted 2023-11-24; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Premature Infant Disease; Newborn Morbidity
Keywords: Newborn; Kangaroo-Mother Care Method; Music Therapy; Intensive Care Units, Neonatal
MeSH Terms: interventions — Music Therapy; Single Person

STUDY DESIGN:
Intervention Model Description: This study adopts a comprehensive approach to explore the effects of three interventions on the well-being and development of newborns in the Neonatal Intensive Care Unit (NICU). The interventions include optimizing the NICU environment for comfort, implementing kangaroo care for parent-infant bonding, and integrating music therapy. The research focuses on two distinct groups within the NICU: premature infants and those undergoing surgical procedures. By examining these interventions across these groups, the study aims to provide nuanced insights into enhancing the holistic care of newborns in critical care settings, tailoring approaches to the unique needs of each population.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kangaroo care (Active Comparator): Kangaroo care Arm subjected to Kangaroo care, a practice involving skin-to-skin contact between the infant and a caregiver.
  Interventions: Other: in the field of rehabilitation and neonatal care: the combination of Kangaroo care method and music therapy
- Music therapy (Active Comparator): Music therapy Arm subjected to music therapy, a practise improving perception of newborns
  Interventions: Other: in the field of rehabilitation and neonatal care: the combination of Kangaroo care method and music therapy

INTERVENTIONS:
Other: in the field of rehabilitation and neonatal care: the combination of Kangaroo care method and music therapy — Kangaroo care is a practice involving skin-to-skin contact between the infant and a caregiver,. Music therapy is a therapeutic approach that utilizes the expressive and emotional qualities of music to address physical, emotional, cognitive needs of individuals.
  Other Names: Kangaroo care method (only); Music therapy (only)

SUMMARY:
Creating a comfortable environment, implementing kangaroo care, and incorporating music therapy are crucial interventions for newborns hospitalized in the Neonatal Intensive Care Unit (NICU). These strategies not only contribute to the physical well-being of the infants but also play a significant role in promoting their emotional and developmental health.

DETAILED DESCRIPTION:
The well-being of newborns in the Neonatal Intensive Care Unit (NICU) is paramount, and establishing a comfortable environment is a fundamental aspect of their care. This involves controlling factors such as temperature, lighting, and noise to mimic the conditions of the womb, creating a soothing and supportive atmosphere for their fragile development. A calm environment is essential for premature infants, as it can contribute to improved weight gain, better sleep patterns, and overall physiological stability.

Kangaroo care, a practice involving skin-to-skin contact between the infant and a caregiver, has proven to be a transformative intervention in NICU settings. This method not only fosters the bond between the baby and their parent but also offers numerous physiological benefits. Kangaroo care has been associated with stabilized heart and respiratory rates, enhanced weight gain, and improved neurodevelopmental outcomes. The close physical contact provides a sense of security and comfort, mimicking the warmth and safety of the mother's womb.

Incorporating music therapy into the care routine of NICU infants has demonstrated positive effects on their well-being. Music has the power to reduce stress, stabilize vital signs, and promote better sleep patterns. Live or recorded lullabies, specifically designed for preterm infants, have been shown to have a calming influence and aid in the regulation of physiological functions. Additionally, music therapy can serve as a valuable tool for parents, offering a means of bonding with their hospitalized newborns and alleviating the stress associated with the NICU experience.

In conclusion, the utility of a comfortable environment, kangaroo care, and music therapy for newborns in the NICU extends beyond basic medical care. These interventions recognize the holistic needs of premature or ill infants, addressing both their physical and emotional requirements. By prioritizing a nurturing and supportive environment, healthcare providers aim to optimize the developmental trajectory of these vulnerable newborns, fostering better outcomes for their long-term health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* newborn hospitalized in NICU

Exclusion Criteria:

* not hospitalized in NICU,
* intubated infants,
* instable clinical condition

Ages: 0 Days to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of kangaroo care and music therapy in premature infants and surgical newborns on weight | from birth to the first 3 years of life
  the effects of kangaroo care and music therapy on anthropometric parameters (weight in grams)
Efficacy of kangaroo care and music therapy in premature infants and surgical newborns on SpO2 | from birth to the first 3 years of life
  the effects of kangaroo care and music therapy on vital signs: saturation in percentage of SpO2
Efficacy of kangaroo care and music therapy in premature infants and surgical newborns on heart rate | from birth to the first 3 years of life
  the effects of kangaroo care and music therapy on vital signs: heart rate in beats for minutes
Efficacy of kangaroo care and music therapy in premature infants and surgical newborns on parenting stress index | from birth to the first 3 years of life
  the effects of kangaroo care and music therapy on scales: Parenting stress index.
  Subscales:1) Parental Distress (PD): personal factors directly related to parenting; 2) Difficult Child (DC): temperament and behavior of the child that influence the parent-child relationship; 3) Parent-Child Dysfunctional Interactions (P-CDI): parent's perception of the child; whether or not expectations are being met, positive behaviors reinforced, etc.
  Assessment Characteristics:36 items Minimum/Maximum Scores: 1) 12 - 60 in each subscale, 2) 36 - 180 total stress score Higher score showed more levels of stress
Efficacy of kangaroo care and music therapy in premature infants and surgical newborns on general movements | from birth to the first 3 years of life
  the effects of kangaroo care and music therapy on scales: General movement optimality scores (GMOS) It differentiated between normal general movements (median 39 [25-75th centile 37-41]), poor repertoire general movements (median 25 [22-29]), cramped-synchronized general movements (median 12 [10-14]).
Efficacy of kangaroo care and music therapy in premature infants and surgical newborns on neurological assessment | from birth to the first 3 years of life
  the effects of kangaroo care and music therapy on scales: Hammersmith Neurological Examination (HNE) HNE assess motor function and overall neurological status. The HNE includes two components: the Hammersmith Functional Motor Scale (HFMS) and the Hammersmith Spinal Muscular Atrophy Functional Rating Scale (HSMARS).
  It is scored on a scale ranging from 0 to 66, with higher scores indicating better motor function.
levels of noise in NICU | from birth to the first 3 years of life
  levels of noise in NICU (assessed as sound pressure levels measured using a dosimeter) in dBA. highter dBA corresponded to more noise

CONTACTS AND LOCATIONS:
Locations (1):
- Neonatal intensive care unit, Catania, Sicily, Italy

IPD SHARING:
Plan to Share IPD: No
newborns meeting predefined inclusion and exclusion criteria will be enrolled to evaluate the impact of environmental noise, kangaroo care, and music therapy during their hospitalization.

REFERENCES:
- [Result] Bieleninik L, Ettenberger M, Epstein S, Elefant C, Arnon S. Potential Psychological and Biological Mechanisms Underlying the Effectiveness of Neonatal Music Therapy during Kangaroo Mother Care for Preterm Infants and Their Parents. Int J Environ Res Public Health. 2021 Aug 13;18(16):8557. doi: 10.3390/ijerph18168557. PMID 34444304